CLINICAL TRIAL: NCT04030715
Title: The Associations Between the Gastric Mucosal Pathology and the Eradication Rate of H.Pylori :A Multicenter Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2018SDU-QILU-G113
Record Dates: First submitted 2019-07-21; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Helicobacter Pylori
Keywords: Gastric Mucosal Pathology; Eradication Rate

STUDY DESIGN:
Intervention Model Description: Use the two-categorical variable , eradicate success or failure ,as a dependent variable, and analyze the influential factors by logistic regression.And then the statistically significant influencing factors like gastric mucosal pathology are obtained.We build a predictive model of the outcome of Hp eradication therapy based on significant influencing factors. The difference with p 0.05 is statistically significant.
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the successful group (Other): divide the subject to two groups based on the success or failure of eradication, and analyze the influential factors of eradication. Build a predictive model for the success of eradication.
  Interventions: Drug: bismuth-containing quadral therapy based on antibiotic susceptibility
- the failure group (Other): divide the subject to two groups based on the success or failure of eradication, and analyze the influential factors of eradication. Build a predictive model for the success of eradication.
  Interventions: Drug: bismuth-containing quadral therapy based on antibiotic susceptibility

INTERVENTIONS:
Drug: bismuth-containing quadral therapy based on antibiotic susceptibility — the different mucosal pathology graded by New Sydney System
  Other Names: gastric mucosal pathology

SUMMARY:
Use the two-categorical variable , eradicate success or failure ,as a dependent variable, and analyze the influential factors by logistic regression.And then the statistically significant influencing factors like gastric mucosal pathology are obtained.We build a predictive model of the outcome of Hp eradication therapy based on significant influencing factors. The difference with p 0.05 is statistically significant.

DETAILED DESCRIPTION:
The subjects who are naiive Hp infection patients recieved the Hp eradication therapy based on antimicrobial susceptibility test.Using success or failure of eradication as a dependent variable, analyze the influential factors by logistic regression.And then the statistically significant influencing factors like gastric mucosal pathology are obtained.We build a predictive model of the outcome of Hp eradication therapy based on significant influencing factors. The difference with p<0.05 is statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged between 18 and 70 years old, with positive H. pylori infection that was not eradicated by previous therapies are included. The H. pylori infection is confirmed by the positive rapid urease test or 13C-breath test.

Exclusion Criteria:

* Patients with significant underlying disease including liver, cardiac, pulmonary, and renal diseases, neoplasia, coagulopathy and genetic diseases, history of gastric surgery, pregnancy, breast-feeding, active gastrointestinal bleeding, patient with peptic ulcer, the use of PPI, NSAID or antibiotics during the 4 weeks prior to enrolment, and previous history of allergic reactions to any of the medications used in this protocol. Patients previously treated with H. pylori eradication regimens or those unwilling to participate in the study were also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Eradication Rate of H.Pylori | 2months
  evaluate the eradication rate of H.Pylori and analysis the association between the gastric mucosal pathology and the eradication rate

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Study Chair — Qilu Hospital of Shandong University; Tian Ma, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China